CLINICAL TRIAL: NCT06113432
Title: CPAP Therapy Through a Helmet or a Full Face Mask in Patients With Acute Hypoxemic Respiratory Failure: a Comparative, Cross-over, Physiological Study
Brief Title: CPAP Therapy Through a Helmet or a Full Face Mask in Patients With Acute Hypoxemic Respiratory Failure: Cross-over Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Helmet-Mask-ARF
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2023-10

CONDITIONS: Pneumonia, Bacterial; Respiratory Failure; COVID-19 Pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial; Respiratory Insufficiency | interventions — Blood Gas Analysis; Respiratory Rate; Heart Rate

STUDY DESIGN:
Intervention Model Description: Enrolled patients will receive all types of respiratory support (helmet CPAP 40 minutes followed by full face mask CPAP 40 minutes or full face mask CPAP 40 minutes followed by helmet CPAP 40 minutes) in a randomized crossover design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Helmet-CPAP then Mask-CPAP (Experimental): CPAP via Helmet 40 minutes, then CPAP via full face mask 40 minutes
  Interventions: Diagnostic Test: Arterial blood gases; Diagnostic Test: Respiratory rate (RR); Diagnostic Test: Pulseoximeter; Diagnostic Test: Assessment of accessory respiratory muscles work; Diagnostic Test: Esophageal pressure measurement; Diagnostic Test: Discomfort Visual Analog Scale (VAS); Diagnostic Test: Noninvasive blood pressure; Diagnostic Test: Heart rate
- Mask-CPAP then Helmet-CPAP (Experimental): CPAP via full face mask 40 minutes, then CPAP via helmet 40 minutes
  Interventions: Diagnostic Test: Arterial blood gases; Diagnostic Test: Respiratory rate (RR); Diagnostic Test: Pulseoximeter; Diagnostic Test: Assessment of accessory respiratory muscles work; Diagnostic Test: Esophageal pressure measurement; Diagnostic Test: Discomfort Visual Analog Scale (VAS); Diagnostic Test: Noninvasive blood pressure; Diagnostic Test: Heart rate

INTERVENTIONS:
Diagnostic Test: Arterial blood gases — Measurement of arterial oxygen and tension and arterial dioxide tension, calculation of arterial partial oxygen tension to inspiratory oxygen fraction (PaO2/FiO2) ratio
Diagnostic Test: Respiratory rate (RR) — Measurement of respiratory rate by waveform analysis using a ventilator
Diagnostic Test: Pulseoximeter — Peripheral capillary oxygen saturation (SpO2) measurement and the ROX-index calculation (SpO2/FiO2/RR)
Diagnostic Test: Assessment of accessory respiratory muscles work — Patrick score calculation. Score: 0. No visible tonic or phasic use of neck muscles. 1. Neck muscles taut but with no respiratory modulation (i.e., tonic activity). 2. Mild respiratory modulation in neck muscle contraction. 3. Moderate phasic activity (no supraclavicular or intercostal indrawing). 4. Vigorous phasic activity with indrawing. 5. Vigorous phasic activity with abdominal paradox.
Diagnostic Test: Esophageal pressure measurement — Esophageal pressure measurement on inspiration and expiration with calculation of delta esophageal pressure, transpulmonary pressure and delta transpulmonary pressure
Diagnostic Test: Discomfort Visual Analog Scale (VAS) — From 1 to 10 points, where 1 point - maximal discomfort, 10 points - minimal discomfort.
Diagnostic Test: Noninvasive blood pressure — Noninvasive blood pressure
Diagnostic Test: Heart rate — Heart rate calculation using electrocardiogram monitoring

SUMMARY:
Observational and randomized trials have demonstrated the high effectiveness of non-invasive helmet ventilatory support, demonstrating a reduction in intubation rate mortality compared with high-flow and standard oxygen therapy. Some pilot physiological studies have shown physiological benefits of helmets compared to the oronasal mask for non-invasive ventilation. The purpose of the study is to compare markers of patient self-inflicted lung injury (P-SILI), patient's comfort, work of breathing, gas exchange, and hemodynamics in patients with acute hypoxemic respiratory failure (AHRF) during non-invasive ventilation (NIV) in continuous positive pressure (CPAP) mode during an oronasal mask ventilation or a combination of a helmet with high-flow oxygenation as an air flow generator.

DETAILED DESCRIPTION:
In December 2019, an outbreak of a novel coronavirus emerged in Wuhan, China and rapidly spread worldwide. The World Health Organization (WHO) declared the outbreak a pandemic on March 11th, 2020. The clinical disease (COVID-19) results in critical illness in about 5% of patients with predominant acute respiratory failure. Observational and randomized trials have demonstrated the high effectiveness of non-invasive helmet ventilatory support, demonstrating a reduction in intubation rate mortality compared with high-flow and standard oxygen therapy. Some pilot physiological studies have shown physiological benefits of helmets compared to the oronasal mask for non-invasive ventilation.

The purpose of the study is to compare markers of patient self-inflicted lung injury (P-SILI) (measuring esophageal pressure, transpulmonary pressure during inspiration and expiration), the patient's work of breathing (assessment of accessory muscles work) patient's comfort by visual-analog scale, gas exchange (by PaO2/FiO2 and Respiration Oxygenation Index (ROX-index), and hemodynamics in patients with acute hypoxemic respiratory failure (AHRF) during non-invasive pulmonary ventilation (NIV) in continuous positive pressure (CPAP) mode during an oronasal mask ventilation or a combination of a helmet with high-flow oxygenation as an air flow generator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute hypoxemic respiratory failure due to community-acquired pneumonia or COVID-19
* The ratio of the partial pressure of oxygen in arterial blood to the inspiratory fraction of oxygen (PaO2/FiO2) is less than 250 mm Hg while breathing atmospheric air
* Respiratory rate more than > 25 per minute.
* Written informed consent

Exclusion Criteria:

* Patients who achieve the following target parameters with only low-flow oxygen therapy (flow up to 15 l/min): SpO2 > 93%, the patient does not have a subjective feeling of fatigue, there is no visible work of the auxiliary respiratory muscles of the neck,
* Unstable hemodynamics (systolic blood pressure <90 mm Hg or mean arterial pressure <65 mm Hg) and/or lactic acidosis (lactate >5 mmol/l and/or clinically diagnosed shock) and/or life-threatening arrhythmia,
* Metabolic acidosis (pH <7.30);
* Patients who were in the ICU for less than 24 hours for any reason
* Primary or secondary lung diseases (exacerbation of chronic obstructive pulmonary disease (COPD), bronchial asthma, interstitial lung diseases, metastatic lung disease)
* Cardiogenic pulmonary edema,
* Chronic diseases in the stag e of decompensation with the development of extrapulmonary organ dysfunction (liver cirrhosis, progression of cancer, CHF),
* Glasgow Coma Scale score <14 points,
* Swallowing disorders
* Hypercapnia (PaCO2>45 mmHg),
* The need for urgent tracheal intubation for any reason,
* Recent head surgery or anatomy that prevents the placement of a helmet or full face mask on the patient,
* Pregnancy,
* Inability to cooperate with staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Inspiratory effort | 40 minutes
  Delta esophageal pressure
Inspiratory delta transpulmonary pressure (stress) | 40 minutes
  Inspiratory delta transpulmonary pressure
Expiratory delta transpulmonary pressure | 40 minutes
  Expiratory delta transpulmonary pressure

SECONDARY OUTCOMES:
Oxygenation | 40 minutes
  PaO2/FiO2 calculation
Respiratory rate | 40 minutes
  Measurement of respiratory rate by waveform analysis using a ventilator
ROX index | 40 minutes
  Peripheral capillary oxygen saturation (SpO2) measurement and the ROX-index calculation (SpO2/FiO2/RR)
Patrick's score | 40 minutes
  Patrick's score measurement, minimum 1point, maximum 5 points, higher score means worse outcome. Score: 0. No visible tonic or phasic use of neck muscles. 1. Neck muscles taut but with no respiratory modulation (i.e., tonic activity). 2. Mild respiratory modulation in neck muscle contraction. 3. Moderate phasic activity (no supraclavicular or intercostal indrawing). 4. Vigorous phasic activity with indrawing. 5. Vigorous phasic activity with abdominal paradox.
Discomfort visual analog scale (VAS) | 40 minutes
  Discomfort VAS score calculation, minimum 1point, maximum 10 points, higher score means better outcome
Noninvasive blood pressure | 40 minutes
  Noninvasive blood pressure
Heart rate | 40 minutes
  Heart rate calculation using electrocardiogram monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Andrey I Yaroshetskiy, MD, PhD, ScD, Principal Investigator — Sechenov University
Locations (1):
- City clinical hospital named after F.I.Inozemtsev, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Antonelli M, Conti G, Pelosi P, Gregoretti C, Pennisi MA, Costa R, Severgnini P, Chiaranda M, Proietti R. New treatment of acute hypoxemic respiratory failure: noninvasive pressure support ventilation delivered by helmet--a pilot controlled trial. Crit Care Med. 2002 Mar;30(3):602-8. doi: 10.1097/00003246-200203000-00019. PMID 11990923
- [Result] Patroniti N, Foti G, Manfio A, Coppo A, Bellani G, Pesenti A. Head helmet versus face mask for non-invasive continuous positive airway pressure: a physiological study. Intensive Care Med. 2003 Oct;29(10):1680-7. doi: 10.1007/s00134-003-1931-8. Epub 2003 Aug 28. PMID 14564379
- [Result] Vargas F, Thille A, Lyazidi A, Campo FR, Brochard L. Helmet with specific settings versus facemask for noninvasive ventilation. Crit Care Med. 2009 Jun;37(6):1921-8. doi: 10.1097/CCM.0b013e31819fff93. PMID 19384209
- [Result] Chiumello D, Pelosi P, Carlesso E, Severgnini P, Aspesi M, Gamberoni C, Antonelli M, Conti G, Chiaranda M, Gattinoni L. Noninvasive positive pressure ventilation delivered by helmet vs. standard face mask. Intensive Care Med. 2003 Oct;29(10):1671-9. doi: 10.1007/s00134-003-1825-9. Epub 2003 Jun 12. PMID 12802491
- [Result] Grieco DL, Menga LS, Eleuteri D, Antonelli M. Patient self-inflicted lung injury: implications for acute hypoxemic respiratory failure and ARDS patients on non-invasive support. Minerva Anestesiol. 2019 Sep;85(9):1014-1023. doi: 10.23736/S0375-9393.19.13418-9. Epub 2019 Mar 12. PMID 30871304
- [Result] Saxena A, Nazir N, Pandey R, Gupta S. Comparison of Effect of Non-invasive Ventilation Delivered by Helmet vs Face Mask in Patients with COVID-19 Infection: A Randomized Control Study. Indian J Crit Care Med. 2022 Mar;26(3):282-287. doi: 10.5005/jp-journals-10071-24155. PMID 35519929
- [Result] Grieco DL, Menga LS, Raggi V, Bongiovanni F, Anzellotti GM, Tanzarella ES, Bocci MG, Mercurio G, Dell'Anna AM, Eleuteri D, Bello G, Maviglia R, Conti G, Maggiore SM, Antonelli M. Physiological Comparison of High-Flow Nasal Cannula and Helmet Noninvasive Ventilation in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2020 Feb 1;201(3):303-312. doi: 10.1164/rccm.201904-0841OC. PMID 31687831